CLINICAL TRIAL: NCT02451657
Title: A Multicenter, Longitudinal, Non-drug Study to Assess the Suitability of Neurocognitive Tests and Functioning Scales for the Measurement of Cognitive and Functioning Changes in Children With Down Syndrome
Brief Title: Non-drug Study to Evaluate the Suitability of Neurocognitive Tests and Functioning Scales for the Measurement of Cognitive and Functioning Changes in Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP29589
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention was administered in this study

SUMMARY:
The aim of this study is to assess the suitability of selected scales (floor/ceiling effects, variability, test-retest reliability) to measure cognitive function in children with Down syndrome over 6 months, and to evaluate the influence of covariates such as age, gender or language on these neurocognitive scales.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6 to 11 with diagnosis of Down syndrome (Trisomy 21). Children may have standard trisomy 21, Robertsonian translocation, isochromosome 21 (so called 21q21q Robertsonian translocation), Down syndrome with reciprocal translocation or mosaicism.
* Down syndrome children meeting clinical diagnostic criteria for generalized anxiety disorders, autism spectrum disorder, attention deficit and hyperactivity disorder, can participate in the study provided they are considered clinically stable or on stable medication for at least 8 weeks prior to the baseline visit.
* Parent or legal guardian/representative and caregiver willing to give written informed consent.
* Subjects with sufficient vision and hearing to engage in study evaluations as referred by their parents. Mild hearing loss will be allowed.

Exclusion Criteria:

* Children who may not be able to comply with the protocol or perform the outcome measures due to significant hearing or visual impairment or other issues judged relevant by the investigators
* Significant sleep disruption or moderate to severe untreated obstructive sleep apnea.
* Any condition which would make the individual or the caregiver, in the opinion of the investigator, unsuitable for the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female children, 6 to 11 years of age inclusive, with diagnosis of Down syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Neurocognitive batteries/tests/scales: Suitability for individuals with Down syndrome assessed by number of tests completed/subjects completing, ceiling/floor effect, variance estimate of baseline/change from baseline | approximately 6 months

SECONDARY OUTCOMES:
Test/re-test reliability: Changes in test results over 6 months | approximately 6 months
Influence of age on several neurocognitive tests and functioning scales in the Down syndrome population | approximately 6 months
Correlations between test results on functioning, adaptive behavior and cognition and IQ level | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke Clin Rsch Institute, Durham, North Carolina
- France (4):
  - CHU de Bordeaux Hopital Pellegrin; Service de Genetique Medicale, Bordeaux
  - Groupement Hospitalier Est-Hopital Femme Mere enfant/Hospice civils de lyon, Bron
  - CHU de Montpellier Hopital Arnaud de Villeneuve; de Génétique, Montpellier
  - CHU de Saint Etienne; Service de Génétique, Saint-Etienne
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago (CHUS); Area Asistencial Integrada de Pediatría, Santiago de Compostela, La Coruña
  - IMIM, Human Pharmacology and Clinical Neurosciences,, Barcelona
  - Hospital Infantil Universitario Niño Jesus; Pediatria Social, Madrid